CLINICAL TRIAL: NCT03089242
Title: MicroRNAs in Acute Kidney Injury (MIRAKI) - a Pilotstudy -
Brief Title: MicroRNAs in Acute Kidney Injury
Acronym: MIRAKI
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Anästhesiologie, PD Dr. Timo Brandenburger, Heinrich-Heine University, Duesseldorf
Other Study IDs: 2017024132
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Kidney Injury in Cardiac Surgery - Expression of microRNAs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation of microRNA expression — no intervention

SUMMARY:
Profiling of microRNAs and long noncoding RNAs (lncRNAs) in patients undergoing cardiac surgery. Analysis: Prediction of acute kidney injury by plasma expression profile of microRNAs?

DETAILED DESCRIPTION:
In this pilot study we will include 150 patients undergoing cardiac surgery in a German university hospital. We will profile microRNA expression in plasma and urine before and at several timepoints after surgery. We will use a preselected panel of microRNAs and lncRNAs for analysis. Goal is to identify microRNAs/lncRNAs that are able to predict the occurence of AKI in these patients.

ELIGIBILITY:
Inclusion Criteria:

* cardiac surgery

Exclusion Criteria:

* preexisting chronic kidney injury
* inclusion in another study
* pregnancy
* Kidney transplantation in history
* GFR < 30 ml/min (glomerular filtration rate)
* ECLS therapy (extracorporal life support)

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cardiac surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
acute kidney injury | 1 year
  AKI Stadium II or III following cardiac surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Timo Brandenburger, M.D., Principal Investigator — Klinik für Anästhesiologie, Heinrich-Heine-Universität Düsseldorf
Locations (1):
- Klinik für Anästhesiologie, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No